CLINICAL TRIAL: NCT07121023
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase Ib Clinical Study to Evaluate the Safety, Efficacy and Kinetic Characteristics of TRD205 Tablets for Postoperative Analgesia After Unilateral Hallux Valgus Orthopedic Surgery
Brief Title: To Evaluate the Safety, Efficacy and Kinetic Characteristics of TRD205 Tablets for Postoperative Analgesia After Unilateral Hallux Valgus Orthopedic Surgery
Acronym: TRD205
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Tide Pharmaceutical Co., Ltd (Industry)
Collaborators: Beijing Jishuitan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRD205-I-02
Record Dates: First submitted 2025-07-29; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Analgesia After Unilateral Hallux Valgus Correction Surgery
Keywords: TRD205 、Postoperative analgesia、unilateral hallux valgus correction surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 200mg treatment group (Experimental): Administered orally every 12 hours for a total of four times；Take 400mg tablets for the first time and 200mg each for the other three times.
  Interventions: Drug: TRD205 tablets
- 400mg treatment group (Experimental): Administered orally every 12 hours for a total of four times；Take800mg tablets for the first time and 400mg each for the other three times.
  Interventions: Drug: TRD205 tablets
- 600mg treatment group (Experimental): Administered orally every 12 hours for a total of four times；Take 1200mg tablets for the first time and 600mg each for the other three times.
  Interventions: Drug: TRD205 tablets
- Placebo (Placebo Comparator): Administered orally every 12 hours for a total of four times；Take 6 tablets for the first time and 3 tablets each for the other three times
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TRD205 tablets — Administered orally every 12 hours for a total of four times；Take TRD205 2 tablets and Placebo 4 tablets for the first time ，TRD205 1 tablets and Placebo 2 tablets each for the other three times.
  Arms: 200mg treatment group
Drug: TRD205 tablets — Administered orally every 12 hours for a total of four times；Take TRD205 4 tablets and Placebo 2 tablets for the first time ，TRD205 2 tablets and Placebo 1 tablets each for the other three times.
  Arms: 400mg treatment group
Drug: TRD205 tablets — Administered orally every 12 hours for a total of four times；Take TRD205 6 tablets and Placebo 0 tablets for the first time ，TRD205 3 tablets and Placebo 0 tablets each for the other three times.
  Arms: 600mg treatment group
Drug: Placebo — Administered orally every 12 hours for a total of four times；Take Placebo 6 tablets for the first time ，Placebo 3 tablets each for the other three times.
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled phase Ib study designed to evaluate the safety, efficacy and PK of TRD205 tablets administered orally .

DETAILED DESCRIPTION:
This study used a placebo as a control to explore the safety, efficacy and pharmacokinetic characteristics of multiple administration of TRD205 tablets at different doses for postoperative analgesia after unilateral hallux valgus correction surgery.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand the purpose and significance of this study, voluntarily participate in this study, voluntarily sign the informed consent form, and voluntarily comply with the trial procedures;
* 18 to 75 years of age, male or female;
* 18 kg/m 2 ≤ BMI ≤ 30 kg/m 2 , Include Cut-off value ;
* American Society of Anesthesiologists (ASA) physical status I to II (Appendix) 6 );
* Elective unilateral hallux valgus orthopedic surgery under general anesthesia (distal osteotomy of the first metatarsal, which can be combined with phalangeal osteotomy) , post-op NRS ≥ 4 points at rest within 4h (timed from the completion of the last suture) ;
* Able to understand the study procedures and the use of various scales involved in this study, and able to communicate effectively with the investigators.

Exclusion Criteria:

* Known allergies or contraindications to the investigational drug and other drugs that may be used during the trial, and those who are not suitable for participating in the trial judged by the investigator;
* Before randomization 5 half-lives The following drugs (subject to the actual package insert, with half-life unknown, then washout at 48h) are used internally, including but not limited to: analgesic drugs (except those specified in the protocol), anticonvulsants, sedative and hypnotic drugs (except those specified in the protocol), anxiolytics, antidepressants, CYP3A4 enzyme inhibitors or inducers, etc. See the List of Prohibited Drugs for the specific types;
* Random First 7 days Inner Use of Chinese herbal medicine with clear analgesic effect as assessed by the investigator;
* Patients who cannot take oral drugs after surgery as judged by the investigator ;
* Combining the following:

  5a Subjects with a history of ipsilateral hallux valgus orthopedic surgery; 5b Complicated with other diseases, deformities and traumas of the foot, and unsuitable for participating in this trial as judged by the investigator; 5c Before signing the ICF 3 History of orthopedic surgery for contralateral hallux valgus within a month, and / Or planning to undergo other surgical procedures (e.g., hallux valgus orthopedic surgery, first metatarsophalangeal arthrodesis) at the same time during the trial;
* Concomitant with other pain conditions that may confound the postoperative pain evaluation as judged by the investigator;
* Sitting systolic blood pressure ≤ 90 mmHg , and or sitting diastolic blood pressure ≤ 5 at screening 0 mmHg (does not include abnormalities between admission to the operating room and emergence from anesthesia) The investigator judged that the abnormality was clinically significant;
* Heart rate < 50 beats per minute or heart rate > 100 beats per minute (excluding Admission to the operating room until emergence from anesthesia Period abnormality), and the abnormality is clinically significant as judged by the investigator; or QTcF > 450 ms in males and QTcF > 470 ms in females [calculated by Fridericia's formula: QTcF = QT/(RR0.33)]; or subjects with a history of severe arrhythmia such as type II atrioventricular block or above, or a history of cardiac insufficiency;
* Patients complicated with severe liver, kidney, cardiovascular and cerebrovascular diseases, metabolic system diseases, and should not participate in this trial at the discretion of the investigator;
* Patients with malignant tumor who are not suitable for participating in the study as judged by the investigator ;
* Patients complicated with mental system diseases (such as schizophrenia, depression, etc.), dementia, migraine, history of epilepsy, and unsuitable for participating in the trial judged by the investigator;
* The subject has a history of psychotropic drug and narcotic drug abuse, drug abuse and alcoholism within 1 year prior to randomization, which means he/she drinks on average more than 2 units of alcohol per day (1 unit = 360 mL of beer or 45 mL of 40% liquor or 150 mL of wine);

Laboratory Abnormalities:

* Abnormal blood routine at screening: neutrophil count < 1.5 × 10 9 /L; platelet count < 100 × 10 9 /L; hemoglobin (Hb) < 80 g/L;
* Abnormal liver function in the screening period: ALT and/or AST ≥ 1.5 times the upper limit of normal, or total bilirubin ≥ 1.5 times the upper limit of normal;
* Abnormal renal function in the screening period: serum creatinine (Cr) ≥ 1.5 times of the upper limit of normal and/or dialysis subjects;
* Abnormal coagulation function during screening period: prothrombin time (PT) prolonged by more than 3 seconds and/or activated partial thromboplastin time (APTT) prolonged by more than 10 seconds;
* Syphilis antibody (SyphilisTP) and human immunodeficiency virus antibody (HIV-Ab) test positive at screening Who, in the judgment of the investigator, are not suitable for the trial ;
* Pregnant or lactating women;
* Those who are unwilling or unable to take effective contraceptive measures during the study or 30 times after the study;
* Participated in other drug or device clinical studies (signed ICF and received treatment with investigational drug/device or placebo) within 3 months prior to randomization;
* Other conditions that the investigator considers inappropriate for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-08-26 (Estimated); Primary Completion 2025-12-27 (Estimated); Study Completion 2025-12-27 (Estimated)

PRIMARY OUTCOMES:
Treatment-Related Adverse Events | 5 Days
  Assessment of all AEs, SAEs and TEAEs

SECONDARY OUTCOMES:
Sum of Pain Intensity Differences from hour 0 to hour 48 (SPID48).Resting state in a resting state | Within 48 hours after the first administration
  Pain intensity (PI) was assessed using the 11-point numeric pain rating scale (0-10; 0 equated to no pain, and 10 equated to the worst pain imaginable) at predose and at15min、30min、45min、1h、1.5h、2h、2.5h、3h、4h、5h、6h and 8 h, and then at 4-hour intervals until hour 48.
Peak Plasma Concentration（Cmax） | 5 days
  To evaluate the pharmacokinetic characteristics of multiple administration of TRD205 tablets for postoperative analgesia after unilateral hallux valgus correction surgery
Area under the plasma concentration versus time curve （AUC） | 5 days
  To evaluate the pharmacokinetic characteristics of multiple administration of TRD205 tablets for postoperative analgesia after unilateral hallux valgus correction surgery
time to peak（Tmax） | 5 days
  To evaluate the pharmacokinetic characteristics of multiple administration of TRD205 tablets for postoperative analgesia after unilateral hallux valgus correction surgery
elimination half life（T1/2） | 5 days
  To evaluate the pharmacokinetic characteristics of multiple administration of TRD205 tablets for postoperative analgesia after unilateral hallux valgus correction surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Jishuitan Hosapital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided